CLINICAL TRIAL: NCT00973401
Title: Retinal Function in Relation to Long Term Changes in the Glucose Level
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Stig Holfort, Glostrup Hospital, department of Ophthalmology
Other Study IDs: Holfort
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Infusion Systems

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic individuals
  Interventions: Other: Insulin pump

INTERVENTIONS:
Other: Insulin pump — Patients receive an insulin pump that optimizes their glucose control.

SUMMARY:
The purpose of this study is to measure the amplitude and implicit time of electroretinogram (ERG), darkadaptation and the calibre of retinal vessels before and after optimized medical treatment of diabetic individuals (a lower blood glucose level) over a period of 12 months. Newly diagnosed type 1 and type 2 diabetics as well as dysregulated type 1 and type 2 diabetic individuals will be included. Retinal vessel calibre measurements will be used as an estimation of changes in the retinal perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Dysregulated type 1 diabetic individuals and newly diagnosed type 1 diabetics. Age >17 < 60 years

Exclusion Criteria:

* Test individuals with significant cataract, prior surgery to the eye, diabetic retinopathy, other serious eye disease, hypertension, other serious systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 30 type 1 diabetics without diabetic retinopathy, with dysregulated metabolic status that is to be medically optimized.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Changes in amplitude/implicit times, retinal vessel diameter, dark adaptation and OCT | 1 week, 1 month, 4 months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark